CLINICAL TRIAL: NCT01148212
Title: Safety and Tolerability of Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Ulrich Palm, MD, Ludwig-Maximilian-University Munich
Other Study IDs: 10/2009
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-01

CONDITIONS: Best Comfort and Lowest Skin Irritation

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Testing safety and tolerability of transcranial direct current stimulation (2 mA, 20 minutes) in four different protocols:

saline-soaked sponges electrode with electrode gel tap-water-soaked sponges tap-water-soaked-sponges + sham stimulation

Outcome measures are tolerability (comfort rating questionnaire), impedances, skin elasticity

ELIGIBILITY:
Inclusion Criteria:

* no neurological or psychiatric illness
* written informed consent

Exclusion Criteria:

* dermatologic diseases
* medication with corticoids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Palm, MD, Principal Investigator — Ludwig-Maximilian-University; Frank Padberg, MD, Study Chair — Ludwig-Maximilian-University
Locations (1):
- Ludwig-Maximilian-University, Dept. of Psychiatry, Munich, Germany